CLINICAL TRIAL: NCT01498276
Title: The Role of the Family Genetics Health Educator in Influencing Health Promoting Behaviors
Brief Title: Family Genetics Health Education and Healthy Behaviors
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120023; 12-HG-0023
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-10-28

CONDITIONS: Diabetes; Cancer; Heart Disease
Keywords: FHH (Family Health History); Natural History; Family Health History; Disease Risk Assessment
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms; Heart Diseases; Hypocalciuric hypercalcemia, familial, type 1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General population: Members of the general population
- Members of under-resourced communities: Participants recruited from under-resourced communities in the Washington, DC area AND in the Southeastern US

SUMMARY:
Background:

- Family-based approaches to reduce disease risk and promote healthy behaviors may be better than targeting individuals. Risk assessments based on family health history may help educate families on disease risks and encourage them to change physical activity and food choices. Specifically, researchers want to better understand the role of mothers in teaching healthy behaviors to their families.

Objectives:

* To determine mothers influence on diet and health-related behaviors.
* To study an intervention tool that connects family health history and disease risk.

Eligibility:

- 18 years of age who have at least one child living at home.

Design:

* Participants will complete a survey over the phone. The survey will take 30 to 40 minutes to complete. The survey will collect family health history on heart disease, diabetes, colorectal cancer, and breast cancer.
* Researchers will give participants a Family Health Package (FHP). The FHP will provide information on family health history and disease risk. It will also recommend behaviors that can reduce health risks.
* Two weeks after sending the FHP, participants will complete a phone survey about the FHP materials and their social networks.
* Some participants will be invited to focus groups. The focus groups will explore diet and health behavior. They will look at food purchasing and preparation and meal sharing. The groups will also discuss attitudes toward healthy eating and physical activity. Each focus group will last 1 to 2 hours.
* Participants will be asked to complete an electronic survey regarding participants health status, causal health beliefs, risk perceptions, and intentions to communicate health information.
* Then, participants will have the opportunity to use the electronic version of the FHP, which will assess family health history.
* After using the FHeP, participants will complete a short electronic survey to identify knowledge and understanding gained from the use of the application, changes in communication intentions, and suggestions for improvements to the application.
* Upon completion of the electronic portion of the study, a study team member will conduct a semi-structured interview to allow the participants to qualitatively evaluate their user experience, including satisfaction and usefulness.
* This study process will take approximately 60-90 minutes.

DETAILED DESCRIPTION:
Lifestyle behaviors, such as diet and physical activity, have been linked to the development of a number of diseases, including cancer, diabetes, and heart disease. Adopting a healthy diet and other preventive health practices are effective ways to reduce associated diseases. However, cancer, diabetes, and heart disease are etiologically complex with multiple risk factors (e.g., genetic, environmental, lifestyle) that tend to cluster in families. Thus, families are an important social context for intervention and lifestyle-focused disease prevention. Our previous research indicates that intergenerational encouragement can motivate behavior change and parents and women tend to be natural encouragers of health behaviors. Therefore, a mixed-method pilot study will be conducted to explore how dietary habits and healthy behaviors are transmitted across family generations and the motivational influence of family health history regarding diseases associated with overweight and diet on improving health behaviors. This pilot study will also assess participants comprehension of an intervention tool outlining family health history and disease risk assessment that will be used in a larger intervention study.

Participants for the paper-based Family Health Package (FHP) Evaluation Phase will be recruited from an existing database developed by the Immersive Virtual Environment Testing Area (IVETA) within the Social and Behavioral Research Branch, NHGRI, consisting of mothers in the Washington, DC area, and through local advertisement and posting on clinicaltrials.gov. Participants will complete a survey interview, providing us with a detailed family health history. From this information, we will create a paper-based FHP that will be sent to participants, consisting of a pedigree, disease risk algorithms, and health guidelines. Participants will be invited to complete a follow-up survey interview, and focus groups will be conducted with a subset of participants. Two initial focus groups will provide feedback on the feasibility and acceptability of the FHP materials. After incorporating revisions, an additional focus group will evaluate the FHP materials. All of the focus groups will also explore diet and health behavior through semi-structured questions. Thematic analysis will identify factors such as influences on health behaviors across generations and the potential impact parents have on initiating and maintaining food choices within their household and the influence of their family of origin on these choices. We have completed an evaluation of the FHP within a predominantly under-resourced, African American community. While the FHP was well received, participants suggested a need for an in-person, community-based, family history health education program centered around concepts presented in the FHP. To that end, we will develop and pilot test a health education program to introduce the FHP to the community. Additional evaluations may be conducted, as necessary, to improve the FHP and reach diverse populations.

The paper-based version of the FHP will be translated into an electronic version, the Family Health ePortal (FHeP). Participants for the electronic Family Health ePortal (FHeP) Evaluation Phase will be recruited from the general population through local advertisement and posting on clinicaltrials.gov. Eligible participants will be consented and invited to access the FHeP. The initial FHeP Evaluation Phase participants will access the FHeP individually to provide feedback on the feasibility and acceptability of the FHeP materials through surveys and a semi-structured interview. After incorporating revisions, subsequent participants will be asked to invite their family members to access the FHeP and evaluate the FHeP materials. FHeP participants will provide demographic, diet, and health behavior information through pre- and post-test surveys as well as survey items within the FHeP. Additional evaluation waves may be conducted, as necessary, to improve the FHeP and increase reach to diverse populations.

We anticipate that the outcomes of these evaluations will 1) provide us with an effective intervention tool for health education and minimizing disease risk within the family, and 2) inform future intervention research. Further study can be directed toward providing family members with appropriate tools to act as family genetic health educators in order to disseminate disease risk information and encourage health promoting behaviors.

ELIGIBILITY:
* INCLUSION CRITERIA:

FHP Evaluation Phase

Eligible participants for the FHP Evaluation Phase will be invited to participate in the study if they meet the following criteria:

1. be able to read and speak English
2. age >= 18 years
3. indicate a willingness to participate in a focus group/discussion.

   * The urban FHP evaluation phase (Washington, DC Metro area) also requires participants to have at least one child. (The rural FHP evaluation, Southeastern US, does not.)

This information will be gauged from the IVETA database and/or through the initial recruitment discussion. This inclusion criteria has been established as we are interested in examining health behaviors across generations in an efficient and timely manner through surveys and focus groups. Focus group participants will be recruited from the larger sample of participants completing surveys. Therefore, participants will be required to read and speak English as the focus

groups will be conducted in English. As this is a pilot study, it is not feasible to recruit large numbers of participants in order to do the focus groups and provide versions of the survey in alternate languages.

-Those who are adopted will be excluded from the study

FHeP Individual Evaluation Phase

Individual Evaluation

Eligible participants will be invited to participate in the study if they meet the followingcriteria:

1. able to read, write, and speak English,
2. able to visit the Clinical Center on the Bethesda, MD main campus for one visit
3. adult
4. demonstrate basic computer literacy

   * NHGRI employees and those who are adopted will be excluded from the study

Family Evaluation

Eligible participants will be invited to participate in the study if they meet the following criteria:

1. able to read, write, and speak English
2. adult
3. demonstrate basic computer literacy
4. willing to invite at least 2 biological family members to participate

   * Those who are adopted will be excluded from the study

FHP Community-based Education Program

Eligible participants will be invited to participate in the study if they meet the following criteria:

1. able to read, write, and speak English,
2. adult, (greater than or equal to 18 years of age), and
3. indicate a willingness to participate in the study.

   * Those who are adopted will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment strategies vary depending upon the substudy in which we are seeking participation. For example, participants may be recruited from the general population. We also seek to enroll members of under-resourced communities. A database that will assist with recruitment in one substudy includes mothers with young children in the Washington, DC area.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2012-01-03 (Actual)

PRIMARY OUTCOMES:
Participants' comprehension of an intervention tool | interim and end-point
  Participants' comprehension of intervention tool outlining family health history and risk assessment of etiologically complex health conditions (heart disease, diabetes, breast and colorectal cancer)
Intergenerational transfer of diet-related behaviors | interim and end-point
  Intergenerational transfer of diet-related behaviors

SECONDARY OUTCOMES:
Efficacy of utilizing mothers to educate family members of disease risk and motivate healthy behaviors. | interim and end-point
  Efficacy of utilizing mothers to educate family members of disease risk and motivate healthy behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Koehly, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - Georgetown Office of Minority Health, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- [Derived] Koehly LM, Morris BA, Skapinsky K, Goergen A, Ludden A. Evaluation of the Families SHARE workbook: an educational tool outlining disease risk and healthy guidelines to reduce risk of heart disease, diabetes, breast cancer and colorectal cancer. BMC Public Health. 2015 Nov 13;15:1120. doi: 10.1186/s12889-015-2483-x. PMID 26566980
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0023.html